CLINICAL TRIAL: NCT06938100
Title: Genotype, Clinical Features and Imaging of Neuroradiological Abnormalities in CADASIL
Acronym: GENICa
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: GENICa
Record Dates: First submitted 2025-04-03; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: CADASIL; CADASIL (Diagnosis)
Keywords: CADASIL; NOTCH3
MeSH Terms: conditions — CADASIL; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In a subsample of patients will be collected plasma and/ or cells tissue specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The project aims to retrospectively and prospectively analyze a population of CADASIL patients in order to study the natural history of the disease by correlating the symptom spectrum with genetic risk and specific neuroradiological and biological markers

- Stratifying patients according to their disease risk, this could contribute to the discovery of personalized therapeutic targets.

ELIGIBILITY:
Inclusion criteria:

* patients of either sex older than 18 years of age;
* finding of a pathogenic mutation on genetic analysis of NOTCH3;
* in the absence of unambiguous mutation, presence of characteristic deposits (GOM) within small vessels at skin biopsy

Exclusion criteria:

* do not meet the diagnostic criteria of CADASIL;
* are unable to give consent for the study due to aphasic or cognitive impairment or because they are deceased at the time of enrollment and their next of kin refuse to give consent for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with genetically confirmed CADASIL and followed in the Cerebrovascular Diseases Outpatient Clinic of Neurology Unit 9 from 2008 to 2023 will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Deepen the knowledge of the clinical phenotype CADASIL patient | T0- T1 (24 months)
  Each patient with CADASIL will undergo to neuroimaging, correlating it with genotype (NOTCH3 gene mutation search outcome), clinical (e.g., the index event, cerebrovascular risk factors, associated manifestations) and instrumental (radiological) characterization.
Identify potentially reversible risk factors for disease progression | 0-24 months
  At baseline, each patient will undergo collection of demographic and clinical data (e.g., the index event, cerebrovascular risk factors, associated manifestations). Disability will be assessed with the modified Rankin Scale (mRS). Neuropsychological assessment will include administration of the Montreal Cognitive Assesment (MoCA) as a screening test. Some components of executive functions will be assessed by Frontal Assesment Battery (F.A.B) scale as a screening test of executive functions, Trail Making Test (TMT) A and B to assess visual search, psychomotor speed and selective attention (TMT test A) and in addition divided and alternating attention and cognitive flexibility by TMT test B, Attentional Matrices to assess sustained attention and visual search and Modified Five Point Test to assess spatial fluency. Finally by means of the Forward Word Span and Backward Digit Span, Verbal Short-Term Memory and Working Memory will be assessed. Alongside the neuropsychological assessment of

SECONDARY OUTCOMES:
Identify clinical, genetic, biological and neuroradiological markers | 0-30 months
  Patients will undergo an MRI study with high-field (3T) equipment consisting of standard morphologic sequences (T1 3D TSE, T2 TSE, 3D FLAIR, SWI, DWI) to assess the extent of leukoencephalopathy, its distribution pattern, the presence of gaps and/or recent ischemic lesions in DWI sequences, perivascular spaces, and concomitant microhemorrhages.
  Laboratory approaches aimed at differentiating progenitors of specific cell populations (e.g., endothelial and vascular smooth muscle cells) from peripheral blood mononuclear cells (PBMCs) or fibroblasts from skin will be performed. In addition, it will be possible to isolate from peripheral blood the plasma component, intended for research and characterization of potential circulating biomarkers, by appropriate multi-omics approaches (transcriptomics, proteomics, lipidomics).
Deepen knowledge of the neuroradiological phenotype of CADASIL patients, depending on the NOTCH3 mutation locus identified (high, moderate or low risk) | 0-30 months
  Patients will undergo an MRI study with high-field (3T), in particular, high-resolution volumetric FLAIR sequences will be used to allow subsequent segmentation analyses of vascular lesions and a more correct quantitative assessment of cortical thickness values of brain areas. Advanced imaging sequences, particularly epi bold resting state for the study of functional brain connectivity, will also be provided.

CONTACTS AND LOCATIONS:
Locations (2):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy
- Hospital Universitario de la Princesa, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutten JW, Van Eijsden BJ, Duering M, Jouvent E, Opherk C, Pantoni L, Federico A, Dichgans M, Markus HS, Chabriat H, Lesnik Oberstein SAJ. The effect of NOTCH3 pathogenic variant position on CADASIL disease severity: NOTCH3 EGFr 1-6 pathogenic variant are associated with a more severe phenotype and lower survival compared with EGFr 7-34 pathogenic variant. Genet Med. 2019 Mar;21(3):676-682. doi: 10.1038/s41436-018-0088-3. Epub 2018 Jul 22. PMID 30032161
- [Background] Ruchoux MM, Maurage CA. CADASIL: Cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy. J Neuropathol Exp Neurol. 1997 Sep;56(9):947-64. PMID 9291937
- [Background] Chabriat H, Joutel A, Dichgans M, Tournier-Lasserve E, Bousser MG. Cadasil. Lancet Neurol. 2009 Jul;8(7):643-53. doi: 10.1016/S1474-4422(09)70127-9. PMID 19539236
- [Background] Opherk C, Peters N, Herzog J, Luedtke R, Dichgans M. Long-term prognosis and causes of death in CADASIL: a retrospective study in 411 patients. Brain. 2004 Nov;127(Pt 11):2533-9. doi: 10.1093/brain/awh282. Epub 2004 Sep 13. PMID 15364702